CLINICAL TRIAL: NCT01032031
Title: The Effect of Dietary Bioactive Compounds on Skin Health in Humans in Vivo
Brief Title: The Effect of Green Tea and Vitamin C on Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: University of Leeds (Other); University of Bradford (Other)
Responsible Party: Principal Investigator, Lesley Rhodes, Professor of Experimental Dermatology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BB/G005575/1; UKCRN 6911 (Registry Identifier: UK Clinical Research Network)
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Skin Cancer
Keywords: Green tea; Vitamin C; Ultraviolet radiation; Inflammation; Photoageing
MeSH Terms: conditions — Skin Neoplasms; Inflammation | interventions — Tea; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green tea + vit C high dose (Active Comparator)
  Interventions: Dietary Supplement: Green tea + vitamin C high dose
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Green tea + vitamin C high dose — One green tea capsule (1250mg catechin) and one vitamin C tablet (100mg) daily for 3 months
  Arms: Green tea + vit C high dose
Dietary Supplement: Placebo capsule — One capsule daily for 3 months
  Arms: Placebo

SUMMARY:
There is little information on the effect of oral bioactive compounds on human skin clinically despite evidence of a beneficial effect from laboratory studies. The aim of this study is to examine the effect of oral bioactive compounds (green tea and vitamin C) on the health of human skin by measuring markers of skin health directly and skin nutrient uptake.

DETAILED DESCRIPTION:
There is little information on the effect of oral catechin, a nutritionally relevant bioactive compound, on skin health in humans in vivo despite considerable evidence for protective effects in experimental studies. Vitamin C is essential for skin health and stabilises catechins in the gut lumen. Ultraviolet radiation (UVR) in sunlight is a key environmental stressor impacting on skin health. Effects include acute inflammation and longer term photodamage.

OBJECTIVE: To examine the protective effect of catechin and vitamin C on UVR-induced inflammation.

STUDY DESIGN

(1) A double-blind randomised controlled nutritional study in 50 healthy volunteers. Volunteers will receive 3 months dietary supplement with high dose bioactive (n=25),or placebo (n=25).

The aim is to quantify the influence of catechin/vitamin C on:

1. UVR-induced inflammation
2. Leukocyte infiltration
3. Inflammatory mediators
4. Markers of photoageing
5. DNA damage
6. Bioavailability will also be assessed

(2) Bioavailability of catechin and vitamin C in skin and blood. Volunteers will receive active dietary supplement. Blood and urine samples will be taken over a period of 6 hours to determine blood bioavailability. Skin biopsies will also be taken to assess skin bioavailability. Volunteers will then receive 3 months of active dietary supplement followed by repeated sampling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Sun-reactive skin type I / II

Exclusion Criteria:

* History of skin cancer
* History of a photosensitivity disorder
* History of a generalised skin disorder
* Sunbathing (including sunbeds) in the past 3 months
* Pregnancy
* Taking photoactive medicine
* Drink tea > 2 cups/day
* Taking nutritional supplements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in the minimum erythemal dose (MED) of ultraviolet radiation. | 3 months
  The UV minimum erythemal dose (MED) will be determined for each study volunteer before and after nutritional supplementation to examine if the intervention can increase the MED and therefore protect against UV-induced erythema.

SECONDARY OUTCOMES:
Intergroup comparison of inflammatory mediators (cytokines/chemokines) in skin biopsy sections and blister fluid. | 3 months
Intergroup comparison of histological biomarkers (leucocytes, markers of photoageing, DNA damage) in skin biopsy sections. | 3 months
Nutrient (polyphenol) bioavailability in samples of skin, blood and urine. | 3 months
  Bioavailability will be assessed in volunteers participating in both the first (RCT) and second (non-randomised bioavailability) parts of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley E Rhodes, MBBS, MD, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Result] Rhodes LE, Darby G, Massey KA, Clarke KA, Dew TP, Farrar MD, Bennett S, Watson RE, Williamson G, Nicolaou A. Oral green tea catechin metabolites are incorporated into human skin and protect against UV radiation-induced cutaneous inflammation in association with reduced production of pro-inflammatory eicosanoid 12-hydroxyeicosatetraenoic acid. Br J Nutr. 2013 Sep 14;110(5):891-900. doi: 10.1017/S0007114512006071. Epub 2013 Jan 28. PMID 23351338
- [Result] Farrar MD, Nicolaou A, Clarke KA, Mason S, Massey KA, Dew TP, Watson RE, Williamson G, Rhodes LE. A randomized controlled trial of green tea catechins in protection against ultraviolet radiation-induced cutaneous inflammation. Am J Clin Nutr. 2015 Sep;102(3):608-15. doi: 10.3945/ajcn.115.107995. Epub 2015 Jul 15. PMID 26178731
- [Result] Clarke KA, Dew TP, Watson RE, Farrar MD, Osman JE, Nicolaou A, Rhodes LE, Williamson G. Green tea catechins and their metabolites in human skin before and after exposure to ultraviolet radiation. J Nutr Biochem. 2016 Jan;27:203-10. doi: 10.1016/j.jnutbio.2015.09.001. Epub 2015 Sep 12. PMID 26454512
- [Result] Clarke KA, Dew TP, Watson RE, Farrar MD, Bennett S, Nicolaou A, Rhodes LE, Williamson G. High performance liquid chromatography tandem mass spectrometry dual extraction method for identification of green tea catechin metabolites excreted in human urine. J Chromatogr B Analyt Technol Biomed Life Sci. 2014 Dec 1;972:29-37. doi: 10.1016/j.jchromb.2014.09.035. Epub 2014 Sep 30. PMID 25306116